CLINICAL TRIAL: NCT04882085
Title: AN OPEN-LABEL, RANDOMIZED, MULTI-CENTER, ACTIVE-CONTROLLED STUDY TO ESTIMATE THE EFFICACY AND SAFETY OF CEFTAZIDIME-AVIBACTAM (CAZ-AVI) VERSUS BEST AVAILABLE TREATMENT (BAT) IN THE TREATMENT OF INFECTIONS DUE TO CARBAPENEM-RESISTANT GRAM-NEGATIVE PATHOGENS IN CHINESE ADULTS
Brief Title: Efficacy and Safety of CAZ-AVI in the Treatment of Infections Due to Carbapenem-resistant G- Pathogens in Chinese Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3591033
Record Dates: First submitted 2021-04-27; First posted 2021-05-11 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-08

CONDITIONS: Urinary Tract Infection; Acute Pyelonephritis; Hospital Acquired Pneumonia; Ventilator-associated Pneumonia; Bacteremia; Intra-abdominal Infection
MeSH Terms: conditions — Urinary Tract Infections; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Bacteremia; Intraabdominal Infections | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAZ-AVI (Experimental): ceftazidime 2g plus avibactam 0.5g
  Interventions: Drug: Zavicefta, Ceftazidime-Avibactam
- Best Available Treatment (Active Comparator): Based on investigative site practice and local epidemiology and guideline
  Interventions: Drug: Best Available Treatment

INTERVENTIONS:
Drug: Zavicefta, Ceftazidime-Avibactam — CAZ-AVI 2.5 g (2 g ceftazidime + 0.5 g avibactam) administered IV as a 2 hour infusion every 8 hours. Dose adjustments are available for participants with CrCL ≤50 mL/min.
  Arms: CAZ-AVI
Drug: Best Available Treatment — main treatment expected to be used as either monotherapy or in combination are colistin, tigecycline, fosfomycin, amikacin, and meropenem
  Arms: Best Available Treatment

SUMMARY:
This is an open-label, randomized, multi-center, interventional, active-controlled Phase 4 study to evaluate the efficacy and safety of CAZ-AVI versus BAT in the treatment of infected participants with selected infection types (Hospital Acquired Pneumonia [HAP] (including Ventilator-Associated Pneumonia [VAP]); Complicated Urinary-Tract Infection [cUTI]; Complicated Intra-Abdominal Infection [cIAI]; Bloodstream Infection [BSI]) due to carbapenem-resistant Gram-negative pathogens in China.This study will be an estimation study. The statistical inference will be based on point estimate and confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age
* Participant must have a diagnosis of an infection (HAP/VAP, cUTI, cIAI, BSI) due to confirmed carbapenem-resistant aerobic Gram-negative pathogens, requiring administration of IV antibacterial therapy
* Participant who had received appropriate prior empiric antibacterial therapy for a carbapenem-resistant pathogen must meet at least 1 of the following criteria: no or no more than 24h; worsening of objective symptoms or signs after at least 48 hours of antibacterial therapy; no change of objective symptoms or signs after at least 72 hours of antibacterial therapy.
* Capable of giving signed informed consent

Exclusion Criteria:

* Other medical or psychiatric condition may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participant is expected to require more than 21 days of treatment
* Participants who need more than 3 systemic antibiotics as part of best available treatment (BAT)
* Previous administration with an investigational drug within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* Participant is pregnant or breastfeeding.
* Acute Physiology and Chronic Health Evaluation (APACHE) II score >30 or <10 using the most recent available data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- China (36):
  - The First Affiliated Hospital of Bengbu Medical, Bengbu, Anhui
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Chizhou People's Hospital, Chizhou, Anhui
  - Fuyang People's Hospital, Fuyang, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Luoyang Central Hospital, Luoyang, Henan
  - NanYang central hospital, Nanyang, Henan
  - Henan provincial people's hospital, Zhengzhou, Henan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Xinhua Hospital, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Kunming (South Hospital), Kunming, Yunnan
  - The First people's Hospital of Kunming, Kunming, Yunnan
  - The First People's Hospital of Kunming Ganmei Hospital (North Hospital), Kunming, Yunnan
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The 2nd Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Jiangyin People's Hospital, Jiangyin
  - Shanghai Fifth People's Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 participants were screened of which 3 participants failed screening and 1 participant was not randomized in the study. A total of 60 participants were enrolled and randomized in the study.
Groups:
- Ceftazidime-Avibactam: Participants with confirmed carbapenem-resistant Gram-negative pathogens infection received Ceftazidime-Avibactam (CAZ-AVI) 2.5 grams (g) (2 g ceftazidime + 0.5 g avibactam) administered intravenously (IV) as 2-hour infusion every 8 hours (q8h) for 14 days.
- Best Available Treatment: Participants with confirmed carbapenem-resistant Gram-negative pathogens infection received best available treatment (BAT) based on investigative site practice and local epidemiology and guideline for 14 days.
Period: Overall Study
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Started | 31 | 29
Safety Analysis Set | 30 | 29
Completed | 24 | 17
Not Completed | 7 | 12
Not completed — Death | 6 | 9
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Randomized not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who took any study intervention. Participants were analyzed according to the product they actually received.
Groups:
- Ceftazidime-Avibactam: Participants with confirmed carbapenem-resistant Gram-negative pathogens infection received CAZ-AVI 2.5 g (2 g ceftazidime + 0.5 g avibactam) administered IV as 2-hour infusion q8h for 14 days.
- Best Available Treatment: Participants with confirmed carbapenem-resistant Gram-negative pathogens infection received BAT based on investigative site practice and local epidemiology and guideline for 14 days.
- Total: Total of all reporting groups
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 1 | 2 | 3
  45-64 years | 8 | 8 | 16
  Greater than equal to (>=) 65 years | 21 | 19 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 22 | 20 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Cure at Test of Cure (TOC) Visit - Microbiologically Modified Intent-to-Treat (mMITT) Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for the index infection (i.e, complicated intra-abdominal infection [cIAI], complicated urinary-tract infection [cUTI], hospital-acquired pneumonia/ventilator-associated pneumonia [HAP/VAP] or bloodstream infection [BSI]) after study treatment. Also, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. The clinical response was assessed by the independent adjudication committee. 95 percent (%) confidence interval (CI) was calculated using Jeffrey's method.
Time Frame: At TOC visit (From Day 21 up to Day 24)
Population: mMITT analysis set (subset of ITT analysis set) included all participants who met minimum disease requirements and received any amount of study therapy, had at least 1 carbapenem-resistant Gram-negative pathogen in an adequate initial/pre-study culture. Participants with inherently resistant pathogens (monomicrobial infections due to any Acinetobacter species) were excluded from mMITT analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 27 | 27
Percentage of participants | 59.3 [40.6 to 76.1] | 25.9 [12.4 to 44.3]

2. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC Visit - Microbiologically Evaluable (ME) Analysis Set
Description: Clinical cure: improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for index infection (i.e. cIAI, cUTI, HAP/VAP or BSI) after study treatment. Also, for cIAI participants, no unplanned drainage or surgical intervention was necessary since initial procedure. 95% CI based on Jeffrey's method. ME analysis set (sub-set of mMITT): participants who received 3 days of study intervention, or received study intervention for >=48 hours with >= 80% compliance, or for <48 hours before discontinuation due to adverse event, no concomitant antibiotics against baseline carbapenem-resistant gram negative pathogens between first dose and TOC (excluding participants with failed study therapy requiring additional antibiotics), had baseline organisms genetically confirmed by central microbiological testing, no indeterminate clinical outcome at end of treatment (EOT) or TOC visits, no important protocol deviations that affect assessment of efficacy.
Time Frame: At TOC visit (From Day 21 up to Day 24)
Population: ME analysis set was evaluated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 14 | 19
Percentage of participants | 78.6 [53.1 to 93.6] | 26.3 [10.8 to 48.4]

3. Secondary Outcome: Percentage of Participants With Clinical Cure at End of Treatment (EOT) Visit -mMITT Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for the index infection (i.e., cIAI, cUTI, HAP/VAP or BSI) after study treatment. Also, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. The clinical response was assessed by the independent adjudication committee. 95% CI was calculated using Jeffrey's method.
Time Frame: At EOT visit (up to 24 hours after the last infusion on Day 14)
Population: mMITT analysis set (subset of ITT analysis set) included all participants who met minimum disease requirements and received any amount of study therapy, had at least 1 carbapenem-resistant Gram-negative pathogen in an adequate initial/pre-study culture. Participants with inherently resistant pathogens (monomicrobial infections due to any Acinetobacter species) were excluded from the mMITT analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 27 | 27
Percentage of participants | 66.7 [47.9 to 82.1] | 29.6 [15.1 to 48.2]

4. Secondary Outcome: Percentage of Participants With Clinical Cure at EOT Visit - ME Analysis Set
Description: Clinical cure: improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for index infection (i.e., cIAI, cUTI, HAP/VAP or BSI) after study treatment. Also, for cIAI participants, no unplanned drainage or surgical intervention was necessary since initial procedure. 95% CI based on Jeffrey's method. ME analysis set (sub-set of mMITT): participants who received 3 days of study intervention, or received study intervention for >=48 hours with >= 80% compliance, or for <48 hours before discontinuation due to adverse event, no concomitant antibiotics against baseline carbapenem-resistant gram negative pathogens between first dose and TOC (excluding participants with failed study therapy requiring additional antibiotics), had baseline organisms genetically confirmed by central microbiological testing, no indeterminate clinical outcome at EOT or TOC visits, no important protocol deviations that affect assessment of efficacy.
Time Frame: At EOT visit (up to 24 hours after the last infusion on Day 14)
Population: ME analysis set was evaluated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 14 | 19
Percentage of participants | 78.6 [53.1 to 93.6] | 31.6 [14.4 to 53.9]

5. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at TOC Visit - mMITT Analysis Set
Description: Favorable microbiological response was defined as eradication or presumed eradication. Eradication was defined as absence (or urine quantification <10^3 colony forming units per milliliter [CFU/mL] for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication was defined as repeat culture of specimens were not performed/ clinically indicated in a participant who had a clinical response of cure (specific to cIAI and HAP/VAP participants). 95% CI was calculated using Jeffrey's method.
Time Frame: At TOC visit (From Day 21 up to Day 24)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 27 | 27
Percentage of participants | 59.3 [40.6 to 76.1] | 25.9 [12.4 to 44.3]

6. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at TOC Visit - ME Analysis Set
Description: Favorable microbiological response=eradication: absence (or urine quantification <10^3 CFU/mL for cUTI participants) of causative pathogen from appropriately obtained specimen at site of infection or presumed eradication: repeat culture of specimens were not performed/clinically indicated in participant who had clinical cure (specific to cIAI,HAP/VAP participants). 95% CI was calculated using Jeffrey's method. ME analysis set: participants received 3 days of study intervention,or received study intervention for >= 48 hours with >=80% compliance or for <48 hours before discontinuation due to adverse event, no concomitant antibiotics against baseline carbapenem-resistant gram negative pathogens between first dose and TOC (excluding participants with failed study therapy requiring additional antibiotics), had baseline organisms confirmed by central microbiological testing, no indeterminate clinical outcome at EOT/TOC, no important protocol deviations that affect assessment of efficacy.
Time Frame: At TOC visit (From Day 21 up to Day 24)
Population: ME analysis set was evaluated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 14 | 19
Percentage of participants | 71.4 [45.5 to 89.5] | 31.6 [14.4 to 53.9]

7. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at EOT Visit - mMITT Analysis Set
Description: Favorable microbiological response was defined as eradication or presumed eradication. Eradication was defined as absence (or urine quantification <10^3 CFU/mL for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication was defined as repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure (specific to cIAI and HAP/VAP participants). 95% CI was calculated using Jeffrey's method.
Time Frame: At EOT visit (Up to 24 hours after last infusion on Day 14)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 27 | 27
Percentage of participants | 81.5 [64.1 to 92.6] | 33.3 [17.9 to 52.1]

8. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at EOT Visit - ME Analysis Set
Description: as for outcome 6
Time Frame: At EOT visit (Up to 24 hours after last infusion on Day 14)
Population: ME analysis set was evaluated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 14 | 19
Percentage of participants | 78.6 [53.1 to 93.6] | 42.1 [22.3 to 64.1]

9. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at TOC Visit - mMITT Analysis Set
Description: as for outcome 7
Time Frame: At TOC visit (From Day 21 up to Day 24)
Population: mMITT analysis set: all participants who met minimum disease requirements, received any amount of study therapy, had at least 1 carbapenem-resistant Gram-negative pathogen in an adequate initial/pre-study culture. Participants with inherently resistant pathogens were excluded. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. 'Number Analyzed' =number of participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 27 | 27
Percentage of participants
  Enterococcus Faecium: number analyzed (Participants) | 0 | 1
  Enterococcus Faecium |  | 0 [0.0 to 85.3]
  Escherichia Coli: number analyzed (Participants) | 1 | 0
  Escherichia Coli | 100.0 [14.7 to 100.0] |
  Klebsiella Pneumoniae: number analyzed (Participants) | 19 | 23
  Klebsiella Pneumoniae | 63.2 [40.9 to 81.8] | 30.4 [14.8 to 50.7]
  Pseudomonas Aeruginosa: number analyzed (Participants) | 8 | 4
  Pseudomonas Aeruginosa | 37.5 [11.9 to 70.5] | 0 [0.0 to 44.5]
  Staphylococcus Aureus: number analyzed (Participants) | 1 | 0
  Staphylococcus Aureus | 0 [0.0 to 85.3] |
  Staphylococcus Capitis Subspecies: number analyzed (Participants) | 1 | 0
  Staphylococcus Capitis Subspecies | 100.0 [14.7 to 100.0] |

10. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at EOT Visit - mMITT Analysis Set
Description: as for outcome 7
Time Frame: At EOT visit (Up to 24 hours after last infusion on Day 14)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 27 | 27
Percentage of participants
  Enterococcus Faecium: number analyzed (Participants) | 0 | 1
  Enterococcus Faecium |  | 0 [0.0 to 85.3]
  Escherichia Coli: number analyzed (Participants) | 1 | 0
  Escherichia Coli | 100.0 [14.7 to 100.0] |
  Klebsiella Pneumoniae: number analyzed (Participants) | 19 | 23
  Klebsiella Pneumoniae | 89.5 [70.3 to 97.7] | 39.1 [21.4 to 59.4]
  Pseudomonas Aeruginosa: number analyzed (Participants) | 8 | 4
  Pseudomonas Aeruginosa | 75.0 [40.8 to 94.4] | 0 [0.0 to 44.5]
  Staphylococcus Aureus: number analyzed (Participants) | 1 | 0
  Staphylococcus Aureus | 0 [0.0 to 85.3] |
  Staphylococcus Capitis Subspecies: number analyzed (Participants) | 1 | 0
  Staphylococcus Capitis Subspecies | 100.0 [14.7 to 100.0] |

11. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause Until Day 28
Description: Percentage of participants who died due to any cause up to Day 28 was reported in this outcome measure. The 95% CI was calculated using the Jeffrey's method.
Time Frame: From first dose of study intervention (Day 1) up to Day 28
Population: Intent-to-Treat (ITT) Analysis Set included all participants randomly assigned to study intervention and who took at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 30 | 29
Percentage of participants | 13.3 [4.7 to 28.7] | 13.8 [4.8 to 29.5]

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent adverse event (TEAE) was any AE that started after the study intervention start date and time.
Time Frame: From start of study treatment on Day 1 up to 32 days after the last dose of study intervention (Up to 46 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 30 | 29
Participants | 24 | 26

13. Secondary Outcome: Number of Participants With Discontinuation Due to Adverse Events
Description: Number of participants who discontinued the study due to adverse events were reported in this outcome measure. Discontinuations from study due to TEAEs included all participants with an AE record indicating that the AE caused permanent discontinuation from the study. Permanent discontinuations from any study intervention due to TEAEs included participants with an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study.
Time Frame: From start of study treatment on Day 1 up to 32 days after the last dose of study intervention (Up to 46 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 30 | 29
Participants
  Discontinuations from study due to TEAEs | 0 | 0
  Permanent discontinuations from any study intervention due to TEAEs | 1 | 6

14. Secondary Outcome: Number of Participants With Potentially Clinically Significant Post-baseline Hematology Values
Description: Potentially clinically significant hematology parameters included Hemoglobin (gram/deciliter), Hematocrit (%), Erythrocytes (10^12/Liter [L]): value < 0.8*lower limit of normal (LLN) and change (Chg) > 20% decrease, value > 1.3*upper limit of normal (ULN) and Chg > 30% increase. Platelets (10^9/L): Value < 0.65*LLN and Chg > 50% decrease, Value > 1.5*ULN and Chg > 100% increase. Leukocytes (10^9/L): Value < 0.65*LLN and Chg > 60% decrease, Value > 1.6*ULN and Chg > 100% increase. Lymphocytes (10^9/L): Value < 0.25*LLN and Chg > 75% decrease, Value > 1.5*ULN and Chg > 100% increase. Neutrophils (10^9/L): Value < 0.65*LLN and Chg > 75% decrease, Value > 1.6*ULN and Chg > 100% increase. Basophils (10^9/L), Eosinophils (10^9/L), Monocytes (10^9/L): Value > 4.0*ULN and Chg > 300% increase. Number of participants with potentially clinically significant values for any hematology parameters were reported in this outcome measure.
Time Frame: From first dose of study treatment (Day 1) until TOC (Up to Day 24)
Population: Safety analysis set included all participants who took any study intervention. Participants were analyzed according to the product they actually received. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 29 | 28
Participants | 7 | 13

15. Secondary Outcome: Number of Participants With Potentially Clinically Significant Post-baseline Clinical Chemistry Values
Description: Potentially clinically significant criteria included Bilirubin(mg/dL): >2.0*ULN and Chg >150% increase (inc).Aspartate Aminotransferase,Alanine Aminotransferase(Units/Liter[U/L]):>3.0*ULN and Chg >200% inc.Alkaline Phosphatase(U/L):<0.5*LLN and Chg >80% decrease (dec),> 2.0*ULN and Chg >100% inc.Protein,Albumin(g/dL):<0.5*LLN and Chg >50% dec,>1.5*ULN and Chg >50% inc.Blood Urea Nitrogen(mg/dL):<0.2*LLN and Chg >100% dec, >3.0*ULN and Chg >200% inc.Creatinine(mg/dL):>2.0*ULN and Chg >100% inc.Sodium(milliequivalent[mEq]/L):<0.85*LLN and Chg >10% dec, >1.1*ULN and Chg >10% inc.Potassium,Chloride(mEq/L):<0.8*LLN and Chg >20% dec, >1.2*ULN and Chg >20% inc.Calcium(mg/dL):<0.7*LLN and Chg >30% dec,> 1.3*ULN and Chg >30% inc.Bicarbonate(mEq/L):<0.7*LLN and Chg >40% dec, >1.3*ULN and Chg >40% inc.Glucose(mg/dL):<0.6*LLN and Chg >40% dec, >3.0*ULN and Chg >200% inc.Number of participants with potentially clinically significant values for any clinical chemistry parameters were reported.
Time Frame: From first dose of study treatment (Day 1) until TOC (Up to Day 24)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
Number analyzed (Participants) | 30 | 28
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: From start of study intervention on Day 1 up to 32 days after the last dose of study intervention (up to 46 days)
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in other, or participant may have experienced both serious and non-serious event. All-cause mortality was assessed in ITT analysis set and SAEs and non-SAEs were assessed in safety population.
Arm/Group | Ceftazidime-Avibactam | Best Available Treatment
All-Cause Mortality (participants affected / at risk) | 6/30 | 9/29
Serious Adverse Events (participants affected / at risk) | 7/30 | 11/29
Other Adverse Events (participants affected / at risk) | 17/30 | 18/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime-Avibactam (N=30) | Best Available Treatment (N=29)
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Circulatory collapse (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime-Avibactam (N=30) | Best Available Treatment (N=29)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Pyrexia (General disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Acid base balance abnormal (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 2
Blood potassium decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 2
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT04882085/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT04882085/SAP_001.pdf